CLINICAL TRIAL: NCT02678442
Title: Pilot-Feasibility Trial of EUS Guided Pancreas Fine Needle Core Biopsy for Whole Exome Sequencing and Genomic Profiling
Brief Title: Endoscopic Ultrasound Guided Fine Needle Biopsy (EUS-FNB-SC) Using a Novel Fork Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Michael Wallace, M.D, MPH, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 15-007801
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FNB first, then FNA (Active Comparator): In an endoscopic ultrasound-guided procedure, Shark Core Fine Needle Biopsy (FNB) will be performed first, followed by Fine Needle Aspiration (FNA).
  Interventions: Device: Fine Needle Biopsy (FNB); Device: Fine Needle Aspiration (FNA)
- FNA first, then FNB (Active Comparator): In an endoscopic ultrasound-guided procedure, Fine Needle Aspiration (FNA) will be performed first, followed by Shark Core Fine Needle Biopsy (FNB).
  Interventions: Device: Fine Needle Biopsy (FNB); Device: Fine Needle Aspiration (FNA)

INTERVENTIONS:
Device: Fine Needle Biopsy (FNB) — The Shark Core FNB is an FDA approved device for sampling of submucosal lesions, mediastinal masses, lymph nodes and intraperitoneal masses. FNB will be performed by 22 gauge for pancreas head and by 19 gauge for all the other sites.
  Other Names: Shark Core Fine Needle Biopsy
Device: Fine Needle Aspiration (FNA) — Fine needle aspiration is a type of biopsy procedure. In fine needle aspiration, a thin needle is inserted into an area of abnormal-appearing tissue or body fluid, and histological material is obtained. FNA will be performed with a standard 25g needle in the usual fashion using back and forth passes for 30 seconds.

SUMMARY:
This is a clinical trial to compare two needles used in biopsy techniques to acquire tissue from pancreatic cancer. The hypothesis is that the tissue yield, as measured by tumor DNA and cellular material is superior for Flexible Needle Biopsy (FNB) compared with conventional Fine Needle Aspiration (FNA). Specifically, FNB will increase the proportion of cases in which sufficient DNA is obtained to allow genomic profiling and whole exome sequencing.

DETAILED DESCRIPTION:
This is a single-blinded randomized controlled trial with paired evaluation of conventional FNA needle versus FNB needle stratified by lesion location (pancreas head tumor versus pancreas body/tail). A minimum of 4 passes ( 2 with each needle) will be performed from all the lesions. After each pass of needle, the on-site cytopathologists will evaluate the adequacy and the degree of the pathological changes in the obtained material. Based on the information provided by the onsite cytopathologists, the endosonographer will repeat the FNA until enough histological material is obtained to confirm a diagnosis. Patients will be assessed immediately after procedure and during the first 30 days with a follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients who are 18 years old or older and are referred for the evaluation of pancreatic mass lesion.
* International Normalized Ratio (INR) less than 1.5 and platelet count of more than 50,000.
* Medically stable to undergo sedation for EUS.
* Signed informed consent

Exclusion Criteria:

* Medical condition that preclude the patient from having a therapeutic procedure regardless of the EUS finding
* Pregnant patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-16; Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Wallace, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | FNB First, Then FNA | FNA First, Then FNB
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | FNB First, Then FNA | FNA First, Then FNB
Started | 25 | 25
Completed | 23 | 23
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FNB First, Then FNA | FNA First, Then FNB | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (14.1) | 70 (9.0) | 69 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 22 | 22 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Total DNA Yield of Adenocarcinoma
Description: Total quantity of DNA obtained from first needle pass of adenocarcinoma, measured in ng/µL.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/µL
Arm/Group | Fine Needle Biopsy (FNB) | Fine Needle Aspiration (FNA)
Number analyzed (Participants) | 37 | 37
ng/µL | 5930.10 (881) | 3365.22 (788)
Statistical Analysis 1: Comparison: Fine Needle Biopsy (FNB) vs Fine Needle Aspiration (FNA); Test type: Superiority; p = 0.01, t-test, 2 sided

2. Secondary Outcome: Total Number of Passes Needed to Obtain Adequate Tissue Sample for Cytology/Histology Diagnosis
Description: The total number of passes required to obtain adequate tissue sample for cytology/histology processing and interpretation.
Time Frame: Baseline
Measure: Median (Full Range); unit: needle passes
Arm/Group | Fine Needle Biopsy (FNB) | Fine Needle Aspiration (FNA)
Number analyzed (Participants) | 50 | 50
needle passes | 5 [0 to 5] | 2 [0 to 5]

3. Secondary Outcome: Core Tissue Length
Description: The length of the tissue core sample acquired, on the first needle pass, measured in centimeters.
Time Frame: Baseline
Measure: Median (Full Range); unit: centimeters
Arm/Group | Fine Needle Biopsy (FNB) | Fine Needle Aspiration (FNA)
Number analyzed (Participants) | 50 | 50
centimeters | 6 [0 to 20] | 2 [0 to 7]
Statistical Analysis 1: Comparison: Fine Needle Biopsy (FNB) vs Fine Needle Aspiration (FNA); Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Concentration of DNA Yield of Adenocarcinoma
Description: The concentration of the DNA from the adenocarcinoma on the first needle pass, measured in micrograms per microliter.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Fine Needle Biopsy (FNB) | Fine Needle Aspiration (FNA)
Number analyzed (Participants) | 37 | 37
µg/mL | 65.00 (8.6) | 37.21 (8.3)
Statistical Analysis 1: Comparison: Fine Needle Biopsy (FNB) vs Fine Needle Aspiration (FNA); Test type: Superiority; p = 0.02, t-test, 2 sided

5. Secondary Outcome: Percentage of Tumor Cellularity
Description: Percent of tumor cellularity with first pass of adenocarcinoma
Time Frame: Baseline
Measure: Median (Full Range); unit: percentage of tumor cellularity
Arm/Group | Fine Needle Biopsy (FNB) | Fine Needle Aspiration (FNA)
Number analyzed (Participants) | 50 | 50
percentage of tumor cellularity | 40 [0 to 90] | 10 [0 to 100]
Statistical Analysis 1: Comparison: Fine Needle Biopsy (FNB) vs Fine Needle Aspiration (FNA); Test type: Superiority; p = .001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Total Number of Subjects Where First-pass Biopsy Contained Adequate Material for Cytologic Interpretation
Description: The total number of subjects whose first-pass biopsy contained adequate material for cytologic interpretation, as determined by a cytopathologist.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Fine Needle Biopsy (FNB) | Fine Needle Aspiration (FNA)
Number analyzed (Participants) | 50 | 50
Participants | 3 | 18

7. Secondary Outcome: Total Number of Subjects Where First-pass Biopsy Contained Adequate Material for High Quality Histologic Interpretation
Description: The number of subjects whose first pass biopsy contained adequate material for high quality histologic interpretation, as determined by a cytopathologist. High quality is defined as being greater than 10 power field in length.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Fine Needle Biopsy (FNB) | Fine Needle Aspiration (FNA)
Number analyzed (Participants) | 50 | 50
Participants | 33 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were assessed immediately after the procedure and during the first 30 days with a follow-up telephone call or clinical visit for each subject, for a total of approximately two and a half years.
Arm/Group | Fine Needle Biopsy (FNB) | Fine Needle Aspiration (FNA)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 2/50 | 0/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fine Needle Biopsy (FNB) (N=50) | Fine Needle Aspiration (FNA) (N=50)
Pancreatitis (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT02678442/Prot_SAP_000.pdf